CLINICAL TRIAL: NCT05588635
Title: Association Between Live Birth Rate and Serum Progesterone on Frozen-thawed Embryo Transfer Day: Retrospective Study
Brief Title: Association Between Live Birth Rate and Serum Progesterone During Hormonal Replacement Therapy
Acronym: PROGEVOL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-05Obs-CHRMT
Record Dates: First submitted 2022-10-10; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Hyperstimulation Syndrome; Frozen-thawed Embryo Transfers
Keywords: serum progesterone; frozen-thawed embryo transfer; live birth rate
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With live birth group: patients with live birth following frozen-thawed embryo transfer
  Interventions: Other: Identification of predictive factors
- Without live birth group: patients without live birth following frozen-thawed embryo transfer
  Interventions: Other: Identification of predictive factors

INTERVENTIONS:
Other: Identification of predictive factors — Evaluation of the following variables : mother age (years), father age (years), serum progesterone (ng/ml), mother body mass index (kg/m2), serum Antimüllerian hormone (AMH) (ng/ml), infertility etiology (yes/no): 4 categories: idiopathic etiology, mixed origin infertility, male infertility, female infertility; smoker status among mothers (yes/no).

SUMMARY:
Nowadays, frozen-thawed embryo transfers (FET) are expending. This practice avoids risk of ovarian hyperstimulation syndrome (OHSS), as well as allowing better synchronization between endometrium and embryo, which is fundamental for pregnancy.

There are several FET protocols, including hormonal replacement therapy cycle (HRT), which enable clinicians to adapt the day of embryo transfer.

However, increase in spontaneous miscarriages was observed with this latter protocol compared to fresh embryo transfers and the other endometrial preparations (natural and stimulated), in relation with the lack of physiological corpus luteum.

Then, Clinicians interrogate about measuring serum progesterone in order to adjust their treatment and/or transfer date. Various studies have shown thresholds below and/or above which pregnancy or live birth rate were lowered.

The main objective is to find a serum progesterone threshold on the day of embryo transfer above which live birth rate is increased. The secondary objectives are to analyze the factors associated with increased serum progesterone on the day of transfer, to analyze the miscarriage rate, and impact of change on luteal phase support on day 12.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 43,
* having frozen-thawed single embryo transfer of a day-5 blastocyst with hormonal replacement therapy, with measurement of serum progesterone on the day of transfer

Exclusion Criteria:

* frozen-thawed transfer of a day-2 or -3 or -6 embryo,
* double embryo transfer,
* other protocol than HRT,
* patient without serum progesterone measurement on the day of transfer

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: patient having frozen-thawed single embryo transfer of a day-5 blastocyst with hormonal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Identification of factors on the embryo transfer day that predict live birth after frozen-thawed embryo transfer | On the day of embryo transfer (Day 0)
  The following variables were compared between groups: mother age (years), father age (years), serum progesterone (ng/ml), mother body mass index (kg/m2), serum Antimüllerian hormone (AMH) (ng/ml), infertility etiology (yes/no): 4 categories: idiopathic etiology, mixed origin infertility, male infertility, female infertility; smoker status among mothers (yes/no).

SECONDARY OUTCOMES:
Pregnancy status | 12 days after embryo transfer (Day 12)
  Pregnancy status (yes/no)
Serum progesterone | 12 days after embryo transfer (Day 12)
  Measurement of serum progesterone (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Ariane GOUTALAND, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No